CLINICAL TRIAL: NCT01246453
Title: A Prospective, Randomized, Double Blind, Controlled Trial to Evaluate Efficacy and Security of Intrapleurally Alteplase vs Urokinase for the Treatment of Complicated Parapneumonic Effusion and Pleural Empyema
Brief Title: Efficacy and Security of Intrapleurally Alteplase vs Urokinase for the Treatment of Complicated Parapneumonic Effusion and Empyema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Hospital Universitari Vall d'Hebron Research Institute, Hospital Universitari Vall d'Hebron Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC07/90479
Record Dates: First submitted 2010-11-18; First posted 2010-11-23 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Empyema, Pleural; Pleural Effusion; Pleural Diseases
MeSH Terms: conditions — Empyema, Pleural; Pleural Effusion; Pleural Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- urokinase (Active Comparator)
  Interventions: Drug: Intrapleurally Alteplase vs Intrapleurally Urokinase
- Alteplase (Active Comparator)
  Interventions: Drug: Intrapleurally Alteplase vs Intrapleurally Urokinase

INTERVENTIONS:
Drug: Intrapleurally Alteplase vs Intrapleurally Urokinase — Alteplase 10 mg and urokinase 100000 intrapleurally administered, once daily for three days and if necessary 6 days

SUMMARY:
1. Objectives:

   * Main objective: To evaluate the efficacy and safety of intrapleural alteplase vs urokinase in patients with complex complicated parapneumonic pleural effusion and empyema.
   * To evaluate the pleural and plasmatic levels of the fibrinolytic system markers after the treatment with alteplase vs urokinase
   * To evaluate the safety of alteplase in the treatment of complex complicated parapneumonic pleural effusion and empyema
2. Design: Multicentric, randomized, parallel, controlled and double blind
3. Main variable: Percentage of curation
4. Study population and number of patients: 204 patients with complex complicated parapneumonic pleural effusions and empyema
5. Duration of the treatment: Three days (main variable), and optional three days (secondary variable)

ELIGIBILITY:
Inclusion Criteria:

* Empyema and Complex Complicated Parapneumonic Pleural Effusion

Exclusion Criteria:

* Pregnancy or breastfeeding
* Critically illness
* Systemic anticoagulant treatment
* Coagulation Disorder
* Bronchopleural fistula
* Active bleeding
* Recent punction of noncompressive artery
* Stroke in the last 6 months
* Major intervention o major traumatism in the last 6 weeks
* Hypersensibility to urokinase or alteplase
* Severe Liver or kidney failure
* Inclusion in another interventional study in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2003-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of intrapleural alteplase vs urokinase in patients with complex complicated parapneumonic pleural effusion and empyema during one year of follow-up. | Evaluation at three and 6 days of treatment
  It will be also an evaluation at one month, six months and one year

SECONDARY OUTCOMES:
To evaluate the pleural and plasmatic levels of the fibrinolytic system markers after the treatment with alteplase vs urokinase | Evaluation at three and 6 days of treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital Arnau de Vilanova, Lleida, Catalonia

REFERENCES:
- [Derived] Aleman C, Porcel JM, Alegre J, Ruiz E, Bielsa S, Andreu J, Deu M, Sune P, Martinez-Sogues M, Lopez I, Pallisa E, Schoenenberger JA, Bruno Montoro J, de Sevilla TF. Intrapleural Fibrinolysis with Urokinase Versus Alteplase in Complicated Parapneumonic Pleural Effusions and Empyemas: A Prospective Randomized Study. Lung. 2015 Dec;193(6):993-1000. doi: 10.1007/s00408-015-9807-6. Epub 2015 Sep 30. PMID 26423784